CLINICAL TRIAL: NCT01593579
Title: Autonomic Phenotype Before and After Akt Inhibition: Akt Therapy for Melanoma Sub-study
Brief Title: Autonomic Phenotype Before and After Akt Inhibition
Status: Withdrawn | Type: Observational
Why Stopped: Planned parent study never enrolled
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Satish R. Raj, Assistant Professor, Vanderbilt University
Other Study IDs: 120390; VR3689 (Other: Vanderbilt)
Record Dates: First submitted 2012-05-04; First posted 2012-05-08 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Diagnosis of Melanoma
Keywords: melanoma; autonomic failure; hypotension; akt therapy
MeSH Terms: conditions — Melanoma; Pure Autonomic Failure; Hypotension | interventions — Supine Position

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Melanoma: Patients with Melanoma that are enrolled in a clinical trial at the Vanderbilt Ingram Cancer Center (VICC) including an arm with an oral Akt inhibitor
  Interventions: Behavioral: Autonomic Function Tests; Other: supine and standing catecholamines

INTERVENTIONS:
Behavioral: Autonomic Function Tests — Patients will undergo Autonomic Function testing (AFT) before and 8 hours after Akt Inhibition therapy. AFT includes: Supine & standing heart rate & blood pressure, 10 minute head up tilt, cardiac output, sinus arrhythmia, hyperventilation, sustained handgrip, valsalva manuever, and cold pressor test.
Other: supine and standing catecholamines — patients will have blood drawn from supine and standing catecholamines.

SUMMARY:
Some Akt inhibitors have produced functional cardiovascular effects such as marked hypotension that may limit their clinical benefit. There are no current data on whether this autonomic failure presents in humans at clinically used doses. We will test the hypothesis that Akt inhibition causes an acute decrease in sympathetic tone and lowers blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with melanoma with a BRAF mutation and relapse following therapy with a BRAF inhibitor
* Enrolled in a clinical trial through the Vanderbilt Ingram Cancer Center (VICC) including an arm with an oral Akt inhibitor
* Able and willing to provide informed consent

Exclusion Criteria:

* Factors which in the investigator's opinion would prevent the participant from completing the protocol, including poor compliance during previous studies or an unpredictable schedule
* Unable to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will have a diagnosis of Melanoma and be participating in a clinical trial with an arm using oral Akt therapy. Patients will be recruited from the Vanderbilt Ingram Cancer Center.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2015-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Drop in systolic blood pressure before and after Akt treatment | 8 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States